CLINICAL TRIAL: NCT01307800
Title: A Phase 3, Multicenter, Double-Blind, Placebo-Controlled Study of 3 Doses of LY2140023 Monohydrate in the Acute Treatment of Patients With DSM-IV-TR Schizophrenia
Brief Title: A Study of LY2140023 in Patients With Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision to stop the trial was based on efficacy results in the overall schizophrenia participant population.
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12430; H8Y-MC-HBBN (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; pomaglumetad methionil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 80 milligrams (mg) LY2140023, BID (Experimental): An 80-mg LY2140023 tablet administered orally, twice daily (BID) for 6 weeks. Prior to randomization, participants will complete a 1-week placebo lead-in period, during which time placebo tablets identical to LY2140023 are administered orally, BID.
  Interventions: Drug: LY2140023
- 40 mg LY2140023, BID (Experimental): A 40-mg LY2140023 tablet administered orally, BID for 6 weeks. Prior to randomization, participants will complete a 1-week placebo lead-in period, during which time, placebo tablets identical to LY2140023 are administered orally, BID.
  Interventions: Drug: LY2140023
- 10 mg LY2140023, BID (Experimental): A 10-mg LY2140023 tablet administered orally, BID for 6 weeks. Prior to randomization, participants will complete a 1-week placebo lead-in period, during which time, placebo tablets identical to LY2140023 are administered orally, BID.
  Interventions: Drug: LY2140023
- Placebo (Placebo Comparator): A placebo tablet administered orally, BID for 7 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2140023 — Administered orally
  Other Names: pomaglumetad methionil
  Arms: 10 mg LY2140023, BID; 40 mg LY2140023, BID; 80 milligrams (mg) LY2140023, BID
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether at least 1 dose level of LY2140023 given to acutely ill patients with schizophrenia will demonstrate significantly greater efficacy as compared to placebo.

DETAILED DESCRIPTION:
The primary objective of this study was to test the hypothesis that at least 1 dose level of LY2140023, given orally to patients with schizophrenia at doses of 80 mg twice daily (BID), 40 mg BID, or 10 mg BID, would demonstrate significantly greater efficacy than placebo at Visit 9, as measured by the change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score.

This was a multicenter, randomized, double-blind, parallel, fixed-dose, Phase 3 study in patients with schizophrenia. The study consisted of 3 periods: a screening and antipsychotic taper phase, a 7-day placebo lead-in phase that was blinded to investigators and patients, and a 6-week active treatment phase.

Eligible patients were those for whom a modification of antipsychotic medication was acutely indicated, in the opinion of the investigator. To be included in the study, patients must have experienced an exacerbation of their illness within the 2 weeks prior to study entry, leading to an intensification of the level of psychiatric care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR); and confirmed by the Structured Clinical Interview for DSM-IV-TR (SCID)
* Non pregnant female patients who agree to use acceptable birth control
* Participants must be considered moderately ill in the opinion of the investigator
* Patients in whom a modification of antipsychotic medication or initiation of antipsychotic medication is acutely indicated in the opinion of the investigator
* Willing to participate in a minimum of 2 weeks of inpatient hospitalization
* One year history of Schizophrenia prior to entering the study
* At study entry patients with a history of antipsychotic treatment must have a lifetime history of at least one hospitalization for the treatment of schizophrenia, not including the hospitalization required for study. Patients who have never taken antipsychotic treatment may enter the study even without a history of hospitalization.
* At study entry patients with a history of antipsychotic treatment must have a history of at least one episode of illness exacerbation requiring an intensification of treatment intervention or care in the last 2 years, not including the present episode of illness. Patients who have never taken antipsychotic treatment may enter the study without a past history of illness exacerbation and intensification of treatment in the last 2 years.
* At study entry patients must have experienced an exacerbation of illness within the 2 weeks prior to entering the study, leading to an intensification of psychiatric care in the opinion of the investigator. If exacerbation occurs in patients who are presently hospitalized, the patient must not have been hospitalized longer than 60 days at entry of the study.
* Patients must be considered reliable and have a level of understanding sufficient to perform all tests and examinations required by the protocol, and be willing to perform all study procedures

Exclusion Criteria:

* Patients who have a history of inadequate clinical response to antipsychotic treatment for schizophrenia
* Diagnosis of substance dependence or substance abuse within 6 month of study entry
* Diagnosis of substance-induced psychosis within 7 days of study entry
* Currently enrolled in, or discontinued within 6 months from a clinical trial involving an investigational product or unapproved use of a drug or device
* Participated in any clinical trial with any pharmacological treatment intervention for which they received a study-related medication in the 6 months prior to study entry
* Previously completed or withdrawn from this study, or any other study investigating LY2140023 or any predecessor molecules with glutamatergic activity
* Treatment with clozapine at doses greater than 200 mg daily within 12 months prior to entering the study, or who have received any clozapine at all during the month before study entry
* Patients currently receiving treatment (within 1 dosing interval, minimum of 4 weeks, prior entering the study) with a depot formulation of an antipsychotic medication
* Patients who are currently suicidal
* Females who are pregnant, nursing, or who intend to become pregnant within 30 days of completing the study
* Patients with uncorrected narrow-angle glaucoma, uncontrolled diabetes, certain diseases of the liver, renal insufficiency, uncontrolled thyroid condition or other serious or unstable illnesses
* Have a history of one or more seizures
* Electroconvulsive therapy (ECT) within 3 months of entering the study or who will have ECT at any time during the study
* History of low white blood cell count
* Medical history of Human Immunodeficiency Virus positive (HIV+) status.
* Higher than normal blood prolactin levels
* Abnormal electrocardiogram results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas, United States
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lipetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Voronezh
- Ukraine (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiev
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia

REFERENCES:
- [Derived] Kinon BJ, Millen BA, Zhang L, McKinzie DL. Exploratory analysis for a targeted patient population responsive to the metabotropic glutamate 2/3 receptor agonist pomaglumetad methionil in schizophrenia. Biol Psychiatry. 2015 Dec 1;78(11):754-62. doi: 10.1016/j.biopsych.2015.03.016. Epub 2015 Mar 19. PMID 25890643

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, participants completed a 1-week placebo lead-in period, during which time placebo tablets were administered orally, twice daily (BID). The Participant Flow and results are based on participants, post-randomization.
Groups:
- 80 mg LY2140023, BID: 160 milligrams per day (mg/day) LY2140023: An 80-mg LY2140023 tablet, administered orally, BID for 6 weeks, post-randomization with the exception of the first 3 days of treatment, post-randomization, when a 40-mg LY2140023 tablet was administered orally, BID.
- 40 mg LY2140023, BID: 80 mg/day LY2140023: A 40-mg LY2140023 tablet, administered orally, BID for 6 weeks, post-randomization.
- 10 mg LY2140023, BID: 20 mg/day LY2140023: A 10-mg LY2140023 tablet, administered orally, BID for 6 weeks, post-randomization.
- Placebo: Placebo tablets, identical to LY2140023, administered orally, BID for 6 weeks, post-randomization.
Period: Overall Study
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Started | 111 | 110 | 118 | 228
Received Treatment (Rec'd Tx) | 111 | 110 | 118 | 228
Rec'd Tx, Not a Placebo (PL) Responder | 102 (PL responders had ≥25% improvement in PANSS total score (defined in measure 1) in lead-in period.) | 103 | 112 | 217
Completed | 57 | 45 | 60 | 118
Not Completed | 54 | 65 | 58 | 110
Not completed — Adverse Event | 9 | 8 | 10 | 14
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 5 | 6 | 2 | 8
Not completed — Perceived Lack of Efficacy | 24 | 23 | 20 | 33
Not completed — Protocol Violation | 0 | 3 | 4 | 5
Not completed — Schedule Conflict Prevented Continuation | 0 | 3 | 1 | 2
Not completed — Sponsor Decision | 6 | 9 | 12 | 28
Not completed — Withdrawal by Subject | 10 | 11 | 8 | 15
Not completed — Participant Moved | 0 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: Participants who received at least 1 dose of study drug according to the treatment group to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo | Total
Number analyzed (Participants) | 111 | 110 | 118 | 228 | 567
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.15 (11.43) | 40.23 (11.39) | 39.80 (10.45) | 40.83 (11.19) | 40.56 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 30 | 66 | 157
  Male | 78 | 82 | 88 | 162 | 410
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 18 | 18 | 35 | 82
  Not Hispanic or Latino | 99 | 92 | 99 | 191 | 481
  Unknown or Not Reported | 1 | 0 | 1 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 1 | 4
  Asian | 0 | 1 | 2 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 2
  Black or African American | 57 | 54 | 59 | 115 | 285
  White | 51 | 50 | 52 | 103 | 256
  More than one race | 1 | 4 | 2 | 5 | 12
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Mexico | 3 | 3 | 4 | 9 | 19
  Puerto Rico | 2 | 2 | 1 | 2 | 7
  Romania | 3 | 4 | 5 | 9 | 21
  Russian Federation | 15 | 13 | 17 | 29 | 74
  Ukraine | 0 | 0 | 2 | 1 | 3
  United States | 88 | 88 | 89 | 178 | 443

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS scale assessed participants (pts) for positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consisted of 30 items. Each item was rated from 1 (absence of symptoms) to 7 (symptoms extremely severe). The sum of the 30 items was defined as the PANSS total score and ranged from 30 to 210. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Pts in efficacy-evaluable intent-to-treat (EE-ITT) population (received at least 1 dose of study drug and not placebo lead-in responders) who had baseline and at least 1 post-baseline PANSS total score. Excluded were pts with missing predefined subpopulation data. Placebo lead-in responder had ≥25% PANSS total score improvement in lead-in period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 91 | 96 | 106 | 206
units on a scale | -3.7 (2.1) | -4.8 (2.3) | -5.0 (2.0) | -7.8 (1.6)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.994, Mixed Models Analysis — The comparison between 80 mg LY2140023, BID and placebo was conducted at a 1-sided alpha level of 0.025, with adjustment for multiplicity by applying the Step-down Dunnett procedure; LS mean difference = 4.1, 95% CI 2-sided [-0.5 to 8.8], Standard Error of Mean 2.4
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.973, Mixed Models Analysis — The comparison between 40 mg LY2140023, BID and placebo was conducted at a 1-sided alpha level of 0.025, with adjustment for multiplicity by applying the Step-down Dunnett procedure; LS mean difference = 3.0, 95% CI 2-sided [-1.9 to 7.9], Standard Error of Mean 2.5
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.896, Mixed Models Analysis — The p-value was 1-sided without adjustment for multiplicity; LS mean difference = 2.8, 95% CI 2-sided [-1.6 to 7.2], Standard Error of Mean 2.2

2. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score in a Predefined Subpopulation of Schizophrenia Participants
Description: The PANSS scale assessed participants for positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consisted of 30 items. Each item was rated from 1 (absence of symptoms) to 7 (symptoms extremely severe). The sum of the 30 items was defined as the PANSS total score and ranged from 30 to 210. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, and gender, as well as the continuous fixed covariates of baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: EE-ITT participants (see Outcome Measure 1 for population definition) in the predefined subpopulation who had a baseline and at least 1 post-baseline PANSS total score. The predefined subpopulation excluded non-Hispanic whites (self-reported) who had A/A genotype at the serotonin 2A receptor (HTR2A) single nucleotide polymorphism (SNP), rs7330461.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 75 | 86 | 90 | 168
units on a scale | -3.4 (2.2) | -4.3 (2.2) | -4.8 (2.0) | -7.7 (1.5)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.955, Mixed Models Analysis — The p-value was 1-sided without adjustment for multiplicity; LS mean difference = 4.3, 95% CI 2-sided [-0.7 to 9.3], Standard Error of Mean 2.5
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.912, Mixed Models Analysis — The p-value was 1-sided without adjustment for multiplicity; LS mean difference = 3.4, 95% CI 2-sided [-1.6 to 8.4], Standard Error of Mean 2.5
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.223, Mixed Models Analysis — The p-value was 1-sided without adjustment for multiplicity; LS mean difference = 2.9, 95% CI 2-sided [-1.8 to 7.7], Standard Error of Mean 2.4

3. Secondary Outcome: Change From Baseline in the Personal and Social Performance (PSP) Score
Description: The PSP scale was a 100-point, single item scale that assessed 4 domains of functioning (personal and social relationships, socially useful activities, self-care, and disturbing and aggressive behaviors). PSP scores ranged from 1 (risk of death) to 100 (excellent functioning) in all 4 domain areas. A higher score indicated a better health state. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants (pts) in the EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline and at least 1 post-baseline PSP score. Excluded were pts with missing predefined subpopulation data. Placebo lead-in responders had a ≥25% PANSS total score improvement in the lead-in period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 67 | 67 | 75 | 149
units on a scale | 7.9 (1.4) | 9.6 (1.6) | 7.1 (1.4) | 8.4 (1.1)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.610, Mixed Models Analysis — The p-value was 1-sided without adjustment for multiplicity; LS mean difference = -0.4, 95% CI 2-sided [-3.5 to 2.6], Standard Error of Mean 1.5
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.223, Mixed Models Analysis — The p-value was 1-sided without adjustment for multiplicity; LS mean difference = 1.3, 95% CI 2-sided [-2.0 to 4.6], Standard Error of Mean 1.7
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.414, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = -1.2, 95% CI 2-sided [-4.2 to 1.7], Standard Error of Mean 1.5

4. Secondary Outcome: Change From Baseline in the Personal and Social Performance (PSP) Score in a Predefined Subpopulation
Description: The PSP scale was a 100-point, single item scale that assessed 4 domains of functioning (personal and social relationships, socially useful activities, self-care, and disturbing and aggressive behaviors). PSP scores ranged from 1 (risk of death) to 100 (excellent functioning) in all 4 domain areas. A higher score indicated a better health state. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, and gender, as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: EE-ITT participants (see Outcome Measure 1 for population definition) in the predefined subpopulation who had a baseline and at least 1 post-baseline PSP score. The predefined subpopulation excluded non-Hispanic whites (self-reported) who had A/A genotype at the serotonin 2A receptor (HTR2A) single nucleotide polymorphism (SNP), rs7330461.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 55 | 61 | 64 | 118
units on a scale | 6.7 (1.4) | 8.6 (1.4) | 6.3 (1.3) | 7.1 (1.0)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.603, Mixed Models Analysis — The p-value was 1-sided without adjustment for multiplicity; LS mean difference = -0.4, 95% CI 2-sided [-3.7 to 2.8], Standard Error of Mean 1.6
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.192, Mixed Models Analysis — The p-value was 1-sided without adjustment for multiplicity; LS mean difference = 1.5, 95% CI 2-sided [-1.9 to 4.8], Standard Error of Mean 1.7
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.619, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = -0.8, 95% CI 2-sided [-3.9 to 2.3], Standard Error of Mean 1.6

5. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score in Females
Description: The PANSS scale assessed participants for positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consisted of 30 items. Each item was rated from 1 (absence of symptoms) to 7 (symptoms extremely severe). The sum of the 30 items was defined as the PANSS total score and ranged from 30 to 210. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Female participants (pts) in EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had baseline and at least 1 post-baseline PANSS total score. Excluded were pts with missing predefined subpopulation data. Placebo lead-in responders had ≥25% PANSS total score improvement in lead-in period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 29 | 23 | 29 | 56
units on a scale | 0.8 (3.8) | 0.0 (4.3) | -4.5 (3.5) | -8.7 (2.7)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = 9.5, 95% CI 2-sided [1.4 to 17.6], Standard Error of Mean 4.1
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.061, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = 8.7, 95% CI 2-sided [-0.4 to 17.8], Standard Error of Mean 4.6
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.304, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = 4.2, 95% CI 2-sided [-3.9 to 12.3], Standard Error of Mean 4.1

6. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Subscores
Description: PANSS subscales included the positive, negative, and general psychopathology subscales. PANSS positive and negative subscales assessed participants for 7 symptoms (positive or negative) associated with schizophrenia. Each item was rated from 1 (absence of symptoms) to 7 (symptoms extremely severe). Scores for both subscales ranged from 7 to 49. PANSS general psychopathology subscale assessed participants for 16 items of general psychopathology associated with schizophrenia. Each item was rated from 1 (absence of symptom) to 7 (symptom extremely severe). General psychopathology scores ranged from 16 to 112. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants (pts) in the EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline and at least 1 post-baseline PANSS subscore. Excluded were pts with missing predefined subpopulation data. Placebo lead-in responders had a ≥25% PANSS total score improvement in the lead-in period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 91 | 96 | 106 | 206
units on a scale
  PANSS Positive Subscore | -1.2 (0.7) | -2.3 (0.7) | -2.0 (0.6) | -2.8 (0.5)
  PANSS Negative Subscore | -0.5 (0.7) | 0.2 (0.7) | -0.6 (0.6) | -1.1 (0.5)
  PANSS General Psychopathology Subscore | -1.9 (1.1) | -2.8 (1.2) | -2.7 (1.1) | -4.2 (0.8)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — The comparison between 80 mg LY2140023, BID and placebo for the change from baseline in PANSS positive subscores was 2-sided without adjustment for multiplicity; LS mean difference = 1.6, 95% CI 2-sided [0.1 to 3.1], Standard Error of Mean 0.8
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.616, Mixed Models Analysis — The comparison between 40 mg LY2140023, BID and placebo for change from baseline in PANSS positive subscores was 2-sided without adjustment for multiplicity; LS mean difference = 0.4, 95% CI 2-sided [-1.2 to 2.0], Standard Error of Mean 0.8
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.307, Mixed Models Analysis — The comparison between 10 mg LY2140023, BID and placebo for change from baseline in PANSS positive subscores was 2-sided without adjustment for multiplicity; LS mean difference = 0.7, 95% CI 2-sided [-0.7 to 2.2], Standard Error of Mean 0.7
Statistical Analysis 4: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.382, Mixed Models Analysis — The comparison between 80 mg LY2140023, BID and placebo for the change from baseline in PANSS negative subscores was 2-sided without adjustment for multiplicity; LS mean difference = 0.7, 95% CI 2-sided [-0.8 to 2.1], Standard Error of Mean 0.7
Statistical Analysis 5: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.107, Mixed Models Analysis — The comparison between 40 mg LY2140023, BID and placebo for the change from baseline in PANSS negative subscores was 2-sided without adjustment for multiplicity; LS mean difference = 1.3, 95% CI 2-sided [-0.3 to 2.8], Standard Error of Mean 0.8
Statistical Analysis 6: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.436, Mixed Models Analysis — The comparison between 10 mg LY2140023, BID and placebo for the change from baseline in PANSS negative subscores was 2-sided without adjustment for multiplicity; LS mean difference = 0.6, 95% CI 2-sided [-0.9 to 2.0], Standard Error of Mean 0.7
Statistical Analysis 7: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.073, Mixed Models Analysis — The comparison between 80 mg LY2140023, BID and placebo for the change from baseline in PANSS general psychopathology subscores was 2-sided without adjustment for multiplicity; LS mean difference = 2.3, 95% CI 2-sided [-0.2 to 4.9], Standard Error of Mean 1.3
Statistical Analysis 8: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.280, Mixed Models Analysis — The comparison between 40 mg LY2140023, BID and placebo for the change from baseline in PANSS general psychopathology subscores was 2-sided without adjustment for multiplicity; LS mean difference = 1.5, 95% CI 2-sided [-1.2 to 4.2], Standard Error of Mean 1.4
Statistical Analysis 9: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.209, Mixed Models Analysis — The comparison between 10 mg LY2140023, BID and placebo for the change from baseline in PANSS general psychopathology subscores was 2-sided without adjustment for multiplicity; LS mean difference = 1.6, 95% CI 2-sided [-0.9 to 4.0], Standard Error of Mean 1.3

7. Secondary Outcome: Percentage of Participants Who Are Responders
Description: Response during the treatment period was defined as a ≥30% decrease from baseline in Positive and Negative Syndrome Scale (PANSS) total score. The PANSS scale assessed participants for positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consisted of 30 items. Each item was rated from 1 (absence of symptoms) to 7 (symptoms extremely severe). The sum of the 30 items was defined as the PANSS total score and ranged from 30 to 210.
Time Frame: Baseline, Week 6
Population: Participants in the EE-ITT population (participants who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline and at least 1 post-baseline PANSS total score. Placebo lead-in responders had a ≥25% PANSS total score improvement in the lead-in period; Last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 91 | 97 | 107 | 206
percentage of participants | 3.3 | 7.2 | 7.5 | 8.3
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.137, Fisher Exact — The p-value was 2-sided without adjustment for multiplicity
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.824, Fisher Exact — The p-value was 2-sided without adjustment for multiplicity
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p > 0.999, Fisher Exact — The p-value was 2-sided without adjustment for multiplicity

8. Secondary Outcome: Time to Response
Description: Time to response is the number of days from randomization until a ≥30% decrease from lead-in baseline in Positive and Negative Syndrome Scale (PANSS) total score. Participants who did not have a response were censored. The PANSS scale assessed participants for positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consisted of 30 items. Each item was rated from 1 (absence of symptoms) to 7 (symptoms extremely severe). The sum of the 30 items was defined as the PANSS total score and ranged from 30 to 210.
Time Frame: Baseline up to Week 6
Population: Participants (pts) in the EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline and at least 1 post-baseline PANSS total score. Number of pts censored: 80 mg LY2140023, BID = 88 pts, 40 mg LY2140023, BID = 90 pts, 10 mg LY2140023, BID = 99 pts, and placebo = 189 pts.
Measure: Median (Full Range); unit: days
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 91 | 97 | 107 | 206
days | NA [NA to NA] — The median (full range) for time to response was not calculable because an insufficient number of participants reached the response event by the final time point (Week 6). | NA [NA to NA] — The median (full range) for time to response was not calculable because an insufficient number of participants reached the response event by the final time point (Week 6). | NA [NA to NA] — The median (full range) for time to response was not calculable because an insufficient number of participants reached the response event by the final time point (Week 6). | NA [NA to NA] — The median (full range) for time to response was not calculable because an insufficient number of participants reached the response event by the final time point (Week 6).

9. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Severity (CGI-S) Scale
Description: The CGI-S was a single item scale that measured severity of illness at the time of assessment. Scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants (pts) in the EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline and at least 1 post-baseline CGI-S score. Excluded were pts with missing predefined subpopulation data. Placebo lead-in responders had a ≥25% PANSS total score improvement in the lead-in period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 97 | 100 | 109 | 213
units on a scale | -0.5 (0.1) | -0.6 (0.1) | -0.5 (0.1) | -0.6 (0.1)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.340, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = 0.12, 95% CI 2-sided [-0.13 to 0.38], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.659, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = -0.06, 95% CI 2-sided [-0.33 to 0.21], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.413, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = 0.10, 95% CI 2-sided [-0.14 to 0.35], Standard Error of Mean 0.12

10. Secondary Outcome: Change From Baseline in the 16-Item Negative Symptoms Assessment (NSA-16) Total Score
Description: The NSA-16 scale was used to help clinicians rate behaviors (not psychopathology) commonly associated with negative symptoms of schizophrenia. The scale contained 16 items and each item was rated from 1 (normal behavior) to 6 (extreme, abnormal behavior). The sum of the 16 items was defined as the NSA-16 total score and ranged from 16 to 96. Higher scores indicated a greater severity of illness. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants (pts) in the EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had baseline and at least 1 post-baseline NSA-16 total score. Excluded were pts with missing predefined subpopulation data. Placebo lead-in responders had ≥25% PANSS total score improvement in the lead-in period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 67 | 67 | 74 | 149
units on a scale | -5.5 (1.4) | -7.1 (1.5) | -6.3 (1.3) | -5.4 (1.1)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.910, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = -0.2, 95% CI 2-sided [-3.1 to 2.7], Standard Error of Mean 1.5
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.265, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = -1.8, 95% CI 2-sided [-4.9 to 1.3], Standard Error of Mean 1.6
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.531, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = -0.9, 95% CI 2-sided [-3.7 to 1.9], Standard Error of Mean 1.4

11. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimension (EQ-5D) Questionnaire
Description: The EQ-5D was a generic, multidimensional, health-related, quality-of-life instrument. The overall health state score was self-reported using a visual analogue scale (VAS) from 0 (worst imaginable health state) to 100 (best imaginable health state). The least squares (LS) mean was estimated using an analysis of covariance (ANCOVA) model that included terms for treatment, pooled investigative site, gender, baseline score and predefined subpopulation ('yes/no').
Time Frame: Baseline, Week 6
Population: Participants in the EE-ITT population (participants who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline and at least 1 post-baseline EQ-5D VAS health state score. Excluded were participants with missing predefined subpopulation data; Last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 84 | 76 | 96 | 180
units on a scale | 6.0 (2.5) | 3.5 (2.8) | 8.2 (2.4) | 6.1 (2.0)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.983, ANCOVA — The comparison between 80 mg LY2140023, BID and placebo for the change from baseline in EQ-5D Questionnaire (VAS) was 2-sided without adjustment for multiplicity; LS mean difference = -0.06, 95% CI 2-sided [-5.21 to 5.10], Standard Error of Mean 2.62
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.351, ANCOVA — The comparison between 40 mg LY2140023, BID and placebo for the change from baseline in EQ-5D Questionnaire (VAS) was 2-sided without adjustment for multiplicity; LS mean difference = -2.56, 95% CI 2-sided [-7.94 to 2.83], Standard Error of Mean 2.74
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.403, ANCOVA — The comparison between 10 mg LY2140023, BID and placebo for the change from baseline in EQ-5D Questionnaire (VAS) was 2-sided without adjustment for multiplicity; LS mean difference = 2.12, 95% CI 2-sided [-2.86 to 7.11], Standard Error of Mean 2.54

12. Secondary Outcome: Change From Baseline on Schizophrenia Resource Utilization Module (S-RUM): Emergency Room (ER) Visits and Outpatient Visits
Description: The S-RUM was a 31-item questionnaire to assess the participant's occupation (work and home), living arrangements, encounters with law enforcement, victimization, ER visits, and outpatient medical visits for a specified period of time. Item 1 asked about the number of ER or equivalent facility visits a participant had for psychiatric (psych) illness during the last year [baseline (BL) assessment] or since the last assessment (post-baseline assessment). Item 2 asked about the number of ER or equivalent facility visits a participant had for non-psychiatric (non-psych) illness or injury during the last year (BL assessment) or since the last assessment (post-BL assessment). Item 5 asked about the number of outpatient visits to other physicians (not psychiatrists or dentists) a participant had during the last year (BL assessment) or since the last assessment (post-BL assessment).
Time Frame: Baseline and Week (Wk) 6
Population: Participants (pts) in EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline S-RUM score for ER/facility visits or outpatient visits. Placebo lead-in responders had a ≥25% PANSS total score improvement in the lead-in period; Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 90 | 82 | 102 | 184
visits
  ER/Facility (Psych), BL | 1.4 (1.8) | 1.1 (1.6) | 1.1 (1.8) | 1.3 (2.4)
  ER/Facility (Psych), Wk 6 | 0.1 (0.6) | 0.0 (0.2) | 0.1 (0.5) | 0.0 (0.3)
  ER/Facility (Non-Psych), BL | 0.4 (0.9) | 0.3 (0.8) | 0.5 (1.3) | 0.4 (0.9)
  ER/Facility (Non-Psych), Wk 6 | 0.0 (0.2) | 0.0 (0.1) | 0.0 (0.2) | 0.0 (0.3)
  Outpatient, BL | 2.3 (10.0) | 1.6 (3.2) | 1.6 (3.3) | 1.6 (2.9)
  Outpatient, Wk 6 | 0.1 (0.7) | 0.1 (0.3) | 0.1 (0.5) | 0.2 (0.8)

13. Secondary Outcome: Change From Baseline on Schizophrenia Resource Utilization Module (S-RUM): Sessions With a Psychiatrist
Description: The S-RUM was a 31-item questionnaire to assess the participant's occupation (work and home), living arrangements, encounters with law enforcement, victimization, emergency room (ER) visits, and outpatient medical visits for a specified period of time. Item 4 asked about the number of sessions with a psychiatrist a participant had, that were not part of this study, during the last year (baseline assessment) or since the last assessment (post-baseline assessment).
Time Frame: Baseline and Week 6
Population: Participants (pts) in EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline S-RUM score for sessions with a psychiatrist. Placebo lead-in responders had a ≥25% PANSS total score improvement in the lead-in period; Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 90 | 82 | 102 | 184
sessions
  Sessions at Baseline | 6.7 (6.8) | 7.1 (7.4) | 7.0 (8.3) | 6.7 (9.4)
  Sessions at Week 6 | 0.6 (2.5) | 0.5 (2.1) | 0.6 (2.6) | 0.2 (0.8)

14. Secondary Outcome: Change From Baseline on Subjective Well-Being Under Neuroleptic Treatment Scale - Short Form (SWN-S) Total Score
Description: The SWN-S was a self-rated scale that measured subjective well-being for the previous 7 days. The SWN-S consisted of 20 items each rated using a 6-point scale from 1 (not at all) to 6 (very much). The sum of the 20 items was defined as the SWN-S total score and ranged from 20 to 120, with higher scores indicating better subjective well-being. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants (pts) in the EE-ITT population (pts who received at least 1 dose of study drug and were not placebo lead-in responders) who had a baseline and at least 1 post-baseline SWN-S total score. Excluded were pts with missing predefined subpopulation data. Placebo lead-in responders had ≥25% PANSS total score improvement in the lead-in period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 66 | 65 | 74 | 148
units on a scale | 1.2 (2.3) | 8.6 (2.5) | 5.9 (2.2) | 6.8 (1.7)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = -5.6, 95% CI 2-sided [-10.4 to -0.8], Standard Error of Mean 2.4
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.487, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = 1.8, 95% CI 2-sided [-3.3 to 6.9], Standard Error of Mean 2.6
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.693, Mixed Models Analysis — The p-value was 2-sided without adjustment for multiplicity; LS mean difference = -0.9, 95% CI 2-sided [-5.6 to 3.7], Standard Error of Mean 2.4

15. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Global Score
Description: The BAS was a 4-item instrument that evaluated akathisia associated with the use of antipsychotic medications. Item 4 was the Global Clinical Assessment (global score) and was rated from 0 (absent) to 5 (severe). The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants in the ITT population (participants who received at least 1 dose of study drug according to the treatment group to which they were randomized) who had a baseline and at least 1 post-baseline BAS global score. Excluded were participants with missing predefined subpopulation data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 106 | 107 | 115 | 224
units on a scale | -0.01 (0.04) | -0.4 (0.04) | 0.0 (0.04) | 0.01 (0.03)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.661, Mixed Models Analysis — The comparison between 80 mg LY2140023, BID and placebo was conducted at a 2-sided alpha level of 0.05 without adjustment for multiplicity; LS mean difference = -0.02, 95% CI 2-sided [-0.10 to 0.06], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.201, Mixed Models Analysis — The comparison between 40 mg LY2140023, BID and placebo was conducted at a 2-sided alpha level of 0.05 without adjustment for multiplicity; LS mean difference = -0.06, 95% CI 2-sided [-0.14 to 0.03], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.697, Mixed Models Analysis — The comparison between 10 mg LY2140023, BID and placebo was conducted at a 2-sided alpha level of 0.05 without adjustment for multiplicity; LS mean difference = -0.02, 95% CI 2-sided [-0.09 to 0.06], Standard Error of Mean 0.04

16. Secondary Outcome: Change From Baseline in Simpson-Angus Scale (SAS) Total Score
Description: The SAS was used to measure Parkinsonian-type symptoms in participants exposed to antipsychotics. The scale consisted of 10 items and each item was rated on a 5-point scale from 0 (complete absence of the condition) to 4 (the presence of the condition in extreme form). The sum of the 10 items was defined as the SAS total score and ranged from 0 to 40. Higher scores indicated a greater severity of illness. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants in the ITT population (participants who received at least 1 dose of study drug according to the treatment group to which they were randomized) who had a baseline and at least 1 post-baseline SAS total score. Excluded were participants with missing predefined subpopulation data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 105 | 107 | 115 | 224
units on a scale | -0.06 (0.11) | -0.18 (0.12) | 0.13 (0.11) | -0.11 (0.08)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.694, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]; LS mean difference = 0.05, 95% CI 2-sided [-0.20 to 0.31], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.596, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]; LS mean difference = -0.07, 95% CI 2-sided [-0.34 to 0.20], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.055, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 3]; LS mean difference = 0.24, 95% CI 2-sided [0.00 to 0.49], Standard Error of Mean 0.13

17. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scales (AIMS) 1-7 Total Score
Description: The AIMS was a 12-item scale designed to record the occurrence of abnormal involuntary (dyskinetic) movements. Items 1 to 10 were rated on a 5-point scale from 0 (no dyskinetic movements) to 4 (severe dyskinetic movements). Items 11 and 12 were 'yes/no' questions regarding the dental condition of a participant. The sum of Items 1 through 7 was defined as the AIMS 1-7 total score and ranged from 0 to 28. Higher scores indicated a greater severity of illness. The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants in the ITT population (participants who received at least 1 dose of study drug according to the treatment group to which they were randomized) who had a baseline and at least 1 post-baseline AIMS 1-7 total score. Excluded were participants with missing predefined subpopulation data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 106 | 107 | 115 | 223
units on a scale | -0.09 (0.12) | -0.01 (0.13) | 0.03 (0.11) | -0.10 (0.09)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.929, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]; LS mean difference = 0.01, 95% CI 2-sided [-0.27 to 0.29], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.519, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]; LS mean difference = 0.09, 95% CI 2-sided [-0.19 to 0.38], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.323, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 3]; LS mean difference = 0.13, 95% CI 2-sided [-0.13 to 0.40], Standard Error of Mean 0.14

18. Secondary Outcome: Percentage of Participants With a Change From Baseline in Suicidal Behaviors and Ideations Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captured the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. Suicidal behavior: a "yes" answer to any 1 of 5 suicidal behavior questions (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide). Suicidal ideation: a "yes" answer to any 1 of 5 suicidal ideation questions (wish to be dead, and 4 different categories of active suicidal ideation). The percentage of participants with treatment-emergent suicidal ideation or behavior (with a change from baseline in C-SSRS) was calculated as the number of participants with an increase in suicidal behavior or ideation over lead-in baseline, divided by the total number of participants multiplied by 100.
Time Frame: Baseline up to Week 6
Population: Participants in the ITT population (participants who received at least 1 dose of study drug according to the treatment group to which they were randomized) who had a baseline and at least 1 post-baseline C-SSRS assessment.
Measure: Number; unit: percentage of participants
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 106 | 108 | 116 | 224
percentage of participants
  Treatment-Emergent Suicidal Ideation | 2.8 | 5.6 | 6.0 | 4.0
  Treatment-Emergent Suicidal Behavior | 0.0 | 0.0 | 0.0 | 0.9
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.758, Fisher Exact — The comparison between 80 mg LY2140023, BID and placebo in the percentage of participants with a change from baseline in C-SSRS suicidal ideation was conducted at a 2-sided alpha level of 0.05 without adjustment for multiplicity
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.576, Fisher Exact — The comparison between 40 mg LY2140023, BID and placebo in the percentage of participants with a change from baseline in C-SSRS suicidal ideation was conducted at a 2-sided alpha level of 0.05 without adjustment for multiplicity
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.425, Fisher Exact — The comparison between 10 mg LY2140023, BID and placebo in the percentage of participants with a change from baseline in C-SSRS suicidal ideation was conducted at a 2-sided alpha level of 0.05 without adjustment for multiplicity

19. Secondary Outcome: Number of Participants Who Discontinued
Description: The reasons for study discontinuation are located in the Participant Flow.
Time Frame: Randomization up to Week 6
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 111 | 110 | 118 | 228
participants | 54 | 65 | 58 | 110

20. Secondary Outcome: Time to Discontinuation
Description: The time to discontinuation, due to any reason, was defined as the total number of days between the randomization date and discontinuation date. Participants who completed the study period were censored. The time to discontinuation was analyzed using Kaplan-Meier estimated survival curves.
Time Frame: Randomization up to Week 6
Population: Participants (pts) in the ITT population (pts who received at least 1 dose of study drug according to the treatment group to which they were randomized). Number of pts censored: 80 mg LY2140023, BID = 57 pts, 40 mg LY2140023, BID = 45 pts, 10 mg LY2140023, BID = 60 pts, and placebo = 118 pts.
Measure: Median (Full Range); unit: days
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 111 | 110 | 118 | 228
days | NA [NA to NA] — The median (full range) was not calculable because an insufficient number of participants reached the event by the final time point (Week 6). | NA [NA to NA] — The median (full range) was not calculated because an insufficient number of participants in all treatment arms reached the event by the final time point (Week 6). | NA [NA to NA] — The median (full range) was not calculable because an insufficient number of participants reached the event by the final time point (Week 6). | NA [NA to NA] — The median (full range) was not calculable because an insufficient number of participants reached the event by the final time point (Week 6).

21. Secondary Outcome: Change From Baseline in Prolactin
Time Frame: Baseline, Week 6
Population: Participants in the ITT population (participants who received at least 1 dose of study drug according to the treatment group to which they were randomized) who had a baseline and at least 1 post-baseline prolactin lab result; Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: micrograms per Liter (mcg/L)
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 101 | 99 | 105 | 208
micrograms per Liter (mcg/L) | 0.6 (15.4) | -0.1 (15.1) | 1.9 (12.2) | -0.8 (13.0)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.444, ANOVA — [p-value comment as in outcome 15, analysis 1]; Analysis of variance (ANOVA) model on rank-transformed change
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.799, ANOVA — [p-value comment as in outcome 15, analysis 2]; ANOVA model on rank-transformed change
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.073, ANOVA — [p-value comment as in outcome 15, analysis 3]; ANOVA model on rank-transformed change

22. Secondary Outcome: Change From Baseline in Weight
Description: The least squares (LS) mean was estimated using a mixed-effects model with repeated measures (MMRM) that included the fixed, categorical effects of treatment, pooled investigative site, visit, treatment-by-visit interaction, gender, and predefined subpopulation ('yes/no'), as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 6
Population: Participants in the ITT population (participants who received at least 1 dose of study drug according to the treatment group to which they were randomized) who had their weight measured at baseline and at least 1 post-baseline visit. Excluded were participants with missing predefined subpopulation data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 105 | 107 | 115 | 223
kilograms (kg) | 0.6 (0.4) | 0.6 (0.4) | 0.2 (0.4) | 0.5 (0.3)
Statistical Analysis 1: Comparison: 80 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.761, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]; LS mean difference = 0.14, 95% CI 2-sided [-0.76 to 1.04], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: 40 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.761, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 2]; LS mean difference = 0.14, 95% CI 2-sided [-0.78 to 1.06], Standard Error of Mean 0.47
Statistical Analysis 3: Comparison: 10 mg LY2140023, BID vs Placebo; Test type: Superiority or Other; p = 0.489, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 3]; LS mean difference = -0.31, 95% CI 2-sided [-1.17 to 0.56], Standard Error of Mean 0.44

23. Other Pre Specified Outcome: Serious Adverse Events (SAEs) Which Occurred During 30 Days After Last Dose of Study Drug
Description: SAEs occurring AFTER a participant's last dose of study drug were to be followed for 30 days, regardless of the investigator's opinion of causation. An SAE was any adverse event (AE) that resulted in death, an initial or prolonged inpatient hospitalization (other than that required by protocol), a life-threatening experience with the immediate risk of dying, a persistent or significant disability/incapacity, a congenital anomaly/birth defect, the occurrence of a seizure or seizure-like event, or an event considered significant by the investigator for any reason. SAEs were reported per Medical Dictionary for Regulatory Activities (MedDRA version 15.1) preferred terms. A summary of serious and all other non-serious AEs reported from Baseline up to Week 6 is located in the Reported Adverse Events module.
Time Frame: Last dose (either early discontinuation or Week 6) through 30-day follow-up period
Population: Participants who received at least 1 dose of study drug according to the treatment group to which they were randomized.
Measure: Number; unit: participants
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Number analyzed (Participants) | 111 | 110 | 118 | 228
participants
  Irritability | 0 | 0 | 1 | 0
  Suicidal ideation | 1 | 0 | 0 | 0
  Homicidal ideation | 1 | 0 | 0 | 0
  Acute myocardial infarction (resulted in death) | 0 | 0 | 0 | 1
  Schizophrenia | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Baseline to 30 Days After Last Dose of Study Drug
Arm/Group | 80 mg LY2140023, BID | 40 mg LY2140023, BID | 10 mg LY2140023, BID | Placebo
Serious Adverse Events (participants affected / at risk) | 4/111 | 6/110 | 5/118 | 11/228
Other Adverse Events (participants affected / at risk) | 70/111 | 70/110 | 75/118 | 129/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mg LY2140023, BID (N=111) | 40 mg LY2140023, BID (N=110) | 10 mg LY2140023, BID (N=118) | Placebo (N=228)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stupor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Schizophrenia (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Irritability (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Homocidal ideation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 80 mg LY2140023, BID (N=111) | 40 mg LY2140023, BID (N=110) | 10 mg LY2140023, BID (N=118) | Placebo (N=228)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 8 (8) | 5 (5) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (5) | 9 (10)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (4) | 6 (8)
Nausea (Gastrointestinal disorders) | 9 (9) | 12 (15) | 12 (12) | 10 (10)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (5) | 7 (8) | 6 (8) | 9 (11)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Pain (General disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 4 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 0/33 (0) | 0/28 (0) | 1/30 (1) | 1/66 (1)
Blood creatine phosphokinase increased (Investigations) | 5 (5) | 4 (4) | 5 (5) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (6) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 5 (6) | 6 (6)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 16 (18) | 12 (13) | 11 (12) | 22 (23)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 5 (5)
Tremor (Nervous system disorders) | 2 (11) | 2 (2) | 3 (3) | 5 (5)
Anxiety (Psychiatric disorders) | 3 (3) | 5 (5) | 3 (3) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4) | 8 (9) | 7 (8)
Psychotic disorder (Psychiatric disorders) | 4 (4) | 3 (3) | 2 (2) | 3 (3)
Schizophrenia (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (2) | 4 (4)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/33 (0) | 0/28 (0) | 0/30 (0) | 2/66 (2)
Menorrhagia (Reproductive system and breast disorders) | 0/33 (0) | 1/28 (1) | 0/30 (0) | 0/66 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/33 (0) | 1/28 (1) | 0/30 (0) | 0/66 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/33 (0) | 1/28 (1) | 0/30 (0) | 0/66 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
An interim analysis for futility was planned and conducted, using a pre-defined threshold. Since probability of trial meeting primary efficacy objectives, given available interim data, was below pre-defined level, trial was stopped early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days